CLINICAL TRIAL: NCT06896331
Title: Inside a Neuron - Ex Vivo Evaluation of Cerebral and Cerebellar Neuronal Activity Through Electrophysiological and Imaging Techniques on Human Tissue from Surgical Activity.
Brief Title: Inside a Neuron - Ex Vivo Evaluation of Cerebral and Cerebellar Neuronal Activity.
Acronym: INSANE
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Francesco Guerrini, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: INSANE
Record Dates: First submitted 2025-03-12; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Human Neural Cells Functioning
Keywords: INSANE, neurons, human, glioma, brain, patch-clamp, HD-MEA
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of brain and cerebellum cortex
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Patients subdued to neurosurgical intervention for the removal of brain or cerebellum primary or secondary tumor

SUMMARY:
Understanding the functioning of human neurons has always been a key element, especially with regard to the translation of the inputs they receive into actions that determine human behavior. However, the vast majority of studies have been performed in animal models due to the difficulty in maintaining neuronal functions ex vivo. Recently, techniques have been illustrated that allow us to obtain slices of brain tissue removed during neurosurgical interventions. The patch-clamp and HD-MEA (high density - microelectrodes array) techniques, used until now for animal samples, can allow us to study the functioning of the neural cells that make up these slices. Furthermore, the exploration of the functioning of the aforementioned cells in pathological conditions can open the field for further therapeutic perspectives.

ELIGIBILITY:
Inclusion Criteria:

* patients with a brain/cerebellum primary or secondary tumor for whom at least partial resection has been planned.

Exclusion Criteria:

* patients with a brain/cerebellum primary or secondary tumor for whom a biopsy has been planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a brain/cerebellum primary or secondary tumor.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | Through study completion, an average of 3 years.
  Intrinsic and extrinsic properties of brain and cerebellum neurons in "health" condition. In particular, following element will be measured:
  * cell membrane capacity and resistance;
  * Sodium and Potassium currents;
  * cell firing frequency.

SECONDARY OUTCOMES:
Secondary endpoint | Through study completion, an average of 3 years.
  Intrinsic and extrinsic properties of brain and cerebellum neurons in "pathological" condition.
  In particular, following element will be measured:
  * cell membrane capacity and resistance;
  * Sodium and Potassium currents; - cell firing frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy